CLINICAL TRIAL: NCT04225663
Title: A Meditation Intervention on Subconcussive Head Impacts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00062234
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2022-11

CONDITIONS: Head Injury Trauma
Keywords: SUB-CONCUSSIVE HEAD IMPACTS; MEDITATION; adolescent athletes; young adult athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The Intervention group will receive 30-minute sessions of guided meditation. During meditation, they will lie down with their backs and torsos elevated by a mat/soft blocks. They will undergo guided breath work.
  Interventions: Behavioral: Guided Meditation
- Control group (No Intervention): The Control group will not have intervention. They will have quiet, independent study for 30-minute sessions.

INTERVENTIONS:
Behavioral: Guided Meditation — Participants will meditate in response to the guidance provided by a trained meditation coach in person.
  Arms: Intervention group

SUMMARY:
The purpose of this research is to explore potential methods of rehabilitating changes observed from repetitive head impacts. Participation in this study will involve functional magnetic resonance (fMRI) imaging, aerobic testing, heart rate variability (HRV) wrist monitor, hypercapnia challenge, a meditation rehabilitation intervention, and filling out survey information concerning subjective well-being.

DETAILED DESCRIPTION:
COLLEGE ATHLETES:

At each study visit, participants will undergo an fMRI-cerebrovascular reactivity (CVR) challenge scanning session as well as an aerobic exercise test on a stationary bike. During the CVR-fMRI scan, the participant will wear a mask that will deliver a blend of oxygen and nitrogen at varying amounts while lying in an MRI scanner. During the aerobic stationary bike assessment, the participant will pedal at a steady state against applied resistance for 10 minutes while wearing an ECG heart rate monitor to observe heart rate. A Biostrap heart rate variability (HRV) wrist monitor will be provided which will be worn daily. The data from the monitor, concerning HRV and sleep, will be collected. The participant will answer a brief survey concerning the previous night's sleep. After the conclusion of the sport's season, there will be a follow up scanning session. After the post-season scan, the participant will participate in a breath work meditation intervention over the following two months, twice a week for a 30 minute meditation session.

HIGH SCHOOL ATHLETES:

Participants will be given a Biostrap HRV monitor which will be worn daily. The data from the monitor, concerning HRV and sleep, will be collected. The participant will answer a brief survey concerning the previous night's sleep. High school athletes will be randomized into one of two study groups, the control group or the intervention group. The intervention group will receive guided meditation over 2 months (twice a week for 30 mins each session), and will ride a stationary bike at 3 time points. The control group will proceed about their lives normally.

ELIGIBILITY:
Inclusion Criteria:

* Participants recruited for this study will be comprised of adolescent and young adult athletes (age-range 13-25) engaged in high school or college contact athletics who are enrolled in an ongoing NIH funded study of subconcussive head impact exposure (Whitlow: R01 NS091602), which acquires pre- and post-season MRI scans and cognitive testing.

Exclusion Criteria:

* Athletes will be excluded from the study if they suffer a concussion over the sports season or during the course of the proposed mediation intervention study. Athletes will be excluded if they experience claustrophobia entering an MRI scanner.

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Neuroimaging | Baseline
  Brain structural data will be acquired with Siemens Skyra 3T MRI with 32-channel head coil.
Neuroimaging | 7 months
  Brain structural data will be acquired with Siemens Skyra 3T MRI with 32-channel head coil.

SECONDARY OUTCOMES:
Heart Rate Variability (HRV) | Baseline
  An aerobic bike test will be used to examine HRV. Upon conclusion of the exercise challenge, HRV will be measured using standard methods, During the warm up and test, they will be wearing apical ECG leads to record heart rate activity.
Heart Rate Variability (HRV) | 7 months
  An aerobic bike test will be used to examine HRV. Upon conclusion of the exercise challenge, HRV will be measured using standard methods, During the warm up and test, they will be wearing a Biostrap ECG heart rate monitor to record heart rate activity.
Measurement of Sleep | Baseline
  Sleep data will be acquired with the Biostrap heart rate variability (HRV) wristband. Sleep will be measured in hours per night.
Measurement of Sleep | 7 months
  Sleep data will be acquired with the Biostrap heart rate variability (HRV) wristband. Sleep will be measured in hours per night.
The Fear of Pain Questionnaire-III (FPQ-III) | Baseline
  A 30-item questionnaire used to assess the fear of pain, including Severe Pain, Minor Pain, and Medical Pain subscales. Each item is rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (extreme), and the total score ranges from 30 to 150.
The Fear of Pain Questionnaire-III (FPQ-III) | 7 months
  A 30-item questionnaire used to assess the fear of pain, including Severe Pain, Minor Pain, and Medical Pain subscales. Each item is rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (extreme), and the total score ranges from 30 to 150.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher T Whitlow, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT04225663/ICF_000.pdf